CLINICAL TRIAL: NCT02375308
Title: Efficacy of Activation-focussed Cognitive Treatment of Depression (ACDT) to Hypnotherapeutic Treatment of Depression (HDT) in Mild to Moderate Major Depression
Brief Title: Efficacy of Cognitive Behavioral to Hypnotherapeutic Treatment of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Anil Batra, Efficacy of Activation-focussed Cognitive Treatment of Depression (ACDT) to Hypnotherapeutic Treatment of Depression (HDT) in Mild to Moderate Major Depression, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTubingen
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Major Depressive Disorder
Keywords: Hypnotherapy; Cognitive Behavioral Therapy; Efficacy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypnotherapeutic Treatment (Experimental): HDT (Hypnotherapeutic Treatment of Depression) focuses on the hypnotic activation and strengthening of individual resources, the use of regression techniques to rebuild positive and negative experiences and the development of positive imaginations for the future.
  Interventions: Behavioral: HDT
- Cognitive Behavioral Treatment (Experimental): ACDT (Activation-focussed Cognitive Treatment of Depression) focuses on psychoeducation, behavior activation, the use of cognitive techniques, and the improvement of social skills.
  Interventions: Behavioral: ACDT

INTERVENTIONS:
Behavioral: HDT — 20 sessions, individual psychotherapy
  Other Names: Hypnotherapeutic Treatment of Depression
  Arms: Hypnotherapeutic Treatment
Behavioral: ACDT — 20 sessions, individual psychotherapy
  Other Names: Cognitive Behavioral Therapy (CBT) of Depression
  Arms: Cognitive Behavioral Treatment

SUMMARY:
The purpose of the study is to compare the efficacy of an Hypnotherapeutic Treatment of Depression to Cognitive Behavioral Treatment of Depression in patients with mild to moderate Major Depressive Episodes.

DETAILED DESCRIPTION:
Cognitive Behavioral Therapy (CBT) is considered to be an effective psychological treatment of mild to moderate Major Depressive Episodes. Effective treatments, however, show a reduction of depressive symptoms only up to 50 % (Luty et al., 2007) which is one reason for the modification of the well-established CBT in the last years. Following the 'third wave' approaches of CBT, e.g. Emotion-Focussed Therapy or Mindfulness-Based Cognitive Therapy, techniques like meditation or the use of systemic or Gestalt techniques within CBT has been applied. Within this context, Hypnotherapy-based strategies can also show an improvement of the current state of the art in depression psychotherapy. However, only few studies conducted randomised controlled trials to study the efficacy of hypnosis for depression as e.g. the comparison of cognitive hypnotherapy to CBT-alone (e.g. Alladin and Alibhai, 2007). With the present study, the efficacy of the Hypnotherapeutic Treatment of Depression (HDT) will be compared to the CBT-based Activation-focussed Cognitive Treatment of Depression (ACDT). Both treatments are individually administered and includes 20 sessions. We expect HDT not being inferior to ACDT in the reduction of depressive symptoms after six months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 (Diagnostic and Statistical Manual) criteria for current mild to moderate Major Depressive Episode (MDE)
* Informed consent
* Fluent in German
* Time for weekly therapy sessions
* Stable antidepressant medication since three months

Exclusion Criteria:

* A history of lifetime bipolar disorder, psychotic symptoms
* A diagnosis of a chronic Major Depressive Disorder (total duration of two years and more)
* Fulfilling the DSM-5 criteria for current severe MDE or scores in MADRS >/= 35 or QIDSC16 (Quick Inventory of Depressive Symptomatology) >/= 16
* Remission of current MDE since more than four weeks prior to inclusion assessment
* Acute risk for suicide
* Severe cognitive impairment (confirmed suspicion with Mini-Mental-State-Test > 25)
* A dominating primary diagnosis of another axis I disorder including anxiety disorders (e.g. Panic disorder, Posttraumatic Stress Disorder, Anorexia nervosa, Borderline personality disorder), or any severe substance-related abuse or dependence disorder
* A physical illness which would interfere with regular psychotherapy sessions
* Outpatient psychotherapy during the last 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-04; Primary Completion 2017-07 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Change from Baseline in MADRS to end of treatment (20 sessions in 20-24 weeks)
  Clinician-rating of depressive symptoms, Primary outcome

SECONDARY OUTCOMES:
QIDS: Quick Inventory of Depressive Symptomatology - Clinician Rating (QIDS-C16) | Change from Baseline to end of therapy and follow-ups (six and 12 months after end of treatment)
  Clinician-rating of depressive symptoms
Patient Health Questionnaire (PHQ-9) | Change from Baseline to end of therapy and follow-ups (six and 12 months after end of treatment)
  Self-report of depressive symptoms
Montgomery-Åsberg Depression Rating Scale (MADRS) | six and 12 months after end of treatment
  Incidence of response rate (symptom reduction > 60%)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Batra, Prof., Principal Investigator — University Hospital Tuebingen
Locations (1):
- Prof. Dr. A. Batra/ Dr. Kristina Fuhr, University Department for Psychiatry and Psychotherapie, Tübingen, Germany

REFERENCES:
- [Background] Luty SE, Carter JD, McKenzie JM, Rae AM, Frampton CM, Mulder RT, Joyce PR. Randomised controlled trial of interpersonal psychotherapy and cognitive-behavioural therapy for depression. Br J Psychiatry. 2007 Jun;190:496-502. doi: 10.1192/bjp.bp.106.024729. PMID 17541109
- [Background] Alladin A, Alibhai A. Cognitive hypnotherapy for depression: an empirical investigation. Int J Clin Exp Hypn. 2007 Apr;55(2):147-66. doi: 10.1080/00207140601177897. PMID 17365072
- [Derived] Fuhr K, Meisner C, Batra A. Long-Term Outcomes of Depression Treatment With Hypnotherapy or Cognitive Behavioral Therapy. J Nerv Ment Dis. 2023 Jul 1;211(7):519-524. doi: 10.1097/NMD.0000000000001647. Epub 2023 Mar 15. PMID 36928627
- [Derived] Fuhr K, Werle D, Batra A. How does early symptom change predict subsequent course of depressive symptoms during psychotherapy? Psychol Psychother. 2022 Mar;95(1):137-154. doi: 10.1111/papt.12370. Epub 2021 Oct 21. PMID 34676660
- [Derived] Fuhr K, Schweizer C, Meisner C, Batra A. Efficacy of hypnotherapy compared to cognitive-behavioural therapy for mild-to-moderate depression: study protocol of a randomised-controlled rater-blind trial (WIKI-D). BMJ Open. 2017 Dec 1;7(11):e016978. doi: 10.1136/bmjopen-2017-016978. PMID 29196478